CLINICAL TRIAL: NCT06280105
Title: A Single-arm, Multicenter, Phase II Trial of Cadonilimab Plus Regorafenib in Patients With Hepatocellular Carcinoma Who Progressed on Camrelizumab Combined With Apatinib
Brief Title: A Trial of Cadonilimab Plus Regorafenib in Patients With Hepatocellular Carcinoma Who Failed Camrelizumab Combined With Apatinib
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Meng Chao Hepatobiliary Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Yongyi Zeng, Director, Meng Chao Hepatobiliary Hospital of Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023_148_01
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: cadonilimab (anti PD-1/CTLA-4 bispecific antibody)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cadonilimab+regorafenib (Experimental)
  Interventions: Drug: Cadonilimab+regorafenib

INTERVENTIONS:
Drug: Cadonilimab+regorafenib — cadonilimab: 6mg/kg iv D1 Q2W; regorafenib: 80mg QD oral; Eligible patients will receive cadonilimab combined with regorafenib, until disease progression or intolerable toxicity or death or withdrawal of informed consent, whichever occurred first

SUMMARY:
To evaluate the efficacy and safety of cadonilimab combined with Regorafenib in patients with hepatocellular carcinoma who failed camrelizumab plus apatinib.

ELIGIBILITY:
Inclusion Criteria:

1. Sign a written informed consent form before enrollment;
2. Age >18 years old, both sex;
3. Histological or pathological confirmed intermediate or advanced hepatocellular carcinoma, or patients with cirrhosis who meet the clinical diagnostic criteria for hepatocellular carcinoma of the American Association for the Study of Liver Diseases (AASLD);
4. Have progressed on the combination treatment of camrelizumab and apatinib for HCC
5. Child-Pugh Class A;
6. ECOG PS score: 0~1;
7. At least 1 measurable lesion (RECIST1.1)
8. Expected survival period≥12 weeks
9. The function of vital organs meets the following requirements (excluding the use of any blood components and cell growth factors within 14 days):

1. Blood routine: Neutrophils≥1.5×109/L Platelet count ≥75×109/L Hemoglobin ≥ 90g/L; 2. Liver and kidney function: Serum creatinine (SCr) ≤ 1.5 times the upper limit of normal (ULN) or creatinine clearance ≥ 50 ml/min (Cockcroft-Gault formula); Total bilirubin (TBIL) ≤ 3 times the upper limit of normal (ULN); Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≤ 10 times the upper limit of normal (ULN); urine protein < 2+; if urine protein ≥ 2+, 24-hour urine protein quantification shows that the protein must be ≤ 1g; 10. Normal coagulation function, no active bleeding or thrombosis disease

1. International normalized ratio INR≤1.5×ULN;
2. Partial thromboplastin time APTT≤1.5×ULN;
3. Prothrombin time PT≤1.5×ULN; 11. Non-surgical sterilization or female patients of childbearing age 12. Subjects voluntarily join this study, have good compliance, and cooperate with safety and survival follow-up

Main Exclusion Criteria:

1. Containing components such as fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, and cholangiocarcinoma that have been previously confirmed by histology/cytology;
2. Have a history of hepatic encephalopathy;
3. Have a history of liver transplantation;
4. There is clinically significant pericardial effusion, and there are clinical symptoms of pleural effusion that require drainage;
5. Clinically apparent ascites is defined as meeting the following criteria: ascites can be detected by physical examination during screening or ascites needs to be drained during screening;
6. Simultaneous infection with HBV and HCV (having a history of HCV infection but negative HCV RNA can be considered as not being infected with HCV);
7. Presence of central nervous system metastasis or meningeal metastasis
8. Bleeding from esophageal or gastric varices caused by portal hypertension has occurred within 6 months before the first dose
9. Patients with any bleeding or bleeding event ≥CTCAE grade 3 within 4 weeks before the first dose
10. Arterial and venous thromboembolic events occurred within 6 months before the first dose
11. Uncontrolled high blood pressure
12. Symptomatic congestive heart failure
13. Severe bleeding tendency or coagulation disorder
14. Have a history of gastrointestinal perforation and/or fistula, intestinal obstruction within 6 months before the first dose
15. Active autoimmune disease or a history of autoimmune disease
16. Patients with HIV
17. According to the investigator's judgment, patients with other serious concomitant diseases that endanger the patient's safety or affect the patient's completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-31 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) per RECIST1.1 | Up to two years
  The proportion of all subjects with the best overall response (BOR) as complete remission (CR) or partial remission (PR) according to RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Progression-free survival（PFS） | Up to two years
  PFS was defined as the time from the first dose to the time of the first documented tumor progression (assessed by RECIST1.1 criteria) or the time of death from any cause, whichever occurred first.
Overall survival（OS） | Up to three years
  Defined as the time from the first dose to the death from any cause.
Duration of response (DOR) | Up to two years
  Defined as the time from the first dose to disease progression or death in patients who achieve complete or partial response
Occurence of AE and SAE | Up to two years
  Occurence of Adverse Event (AE) and Serious Adverse Event (SAE) （NCI CTCAE 5.0）

CONTACTS AND LOCATIONS:
Locations (1):
- Mengchao Hepatobiliary Hospital, Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No